CLINICAL TRIAL: NCT06068920
Title: Evaluation of Distress and Related Factors in Patients With Rheumatoid Arthritis
Brief Title: Distress in Rheumatoid Arthritis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Altınay Göksel Karatepe, Professor Doctor, Bozyaka Training and Research Hospital
Other Study IDs: IBEAH
Record Dates: First submitted 2023-09-29; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Arthritis, Rheumatoid; Distress, Emotional
Keywords: rheumatoid arthritis, distress
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Distress evaluation — To evaluate the effects of psychological distress caused by living with a chronic disease such as rheumatoid arthritis.

SUMMARY:
The goal of this observational study is to determine the frequency of psychological distress caused by the rheumatoid arthritis disease in patients with rheumatoid arthritis and to determine the factors associated with the distress.

A routine rheumatoid arthritis patient examination (number of swollen and tender joints, disease activity, functional status, etc.) will be performed by the doctor to evaluate the patients. Patients will be asked to fill out the questionnaires to evaluate their functional status and distress levels.

Demographic data such as age, gender, body mass index and disease duration will be recorded during routine follow-up of the patients. The duration of morning stiffness, the number of swollen and tender joints, disease activity and functional status will be evaluated by the doctor. Disease activity will be evaluated with the DAS 28 score and functional status will be evaluated with the Health Assessment Questionnaire. Rheumatoid Arthritis Distress Scale (RADS) will be used to evaluate the distress due to rheumatoid arthritis.Patients will be asked to fill out the questionnaires to evaluate their functional status and distress levels.

DETAILED DESCRIPTION:
Demographic data such as age, gender, body mass index and disease duration will be recorded during routine follow-up of the patients. The duration of morning stiffness, the number of swollen and tender joints, disease activity and functional status will be evaluated by the doctor. Disease activity will be evaluated with the DAS 28 score and functional status will be evaluated with the Health Assessment Questionnaire. Rheumatoid Arthritis Distress Scale (RADS) will be used to evaluate the distress due to rheumatoid arthritis.

DAS28 score is a score calculated by a mathematical formula based on the patient's swollen and tender joint counts, erythrocyte sedimentation rate and the patient's global assessment of disease activity.

The Health Assessment Questionnaire consists of twenty items and evaluates the degree of difficulty patients have in performing daily living activities. The total score varies between 0 and 3, with a higher score indicating a more serious impact on daily functional status.

Rheumatoid Arthritis Distress Scale (RADS) is a scale developed to evaluate the psychological distress experienced in patients with rheumatoid arthritis due to the effects of the disease. The total score varies between 0 and 5, with a higher score indicating more impact.

ELIGIBILITY:
Inclusion Criteria:

1. Having rheumatoid arthritis over the age of 18
2. Having the cognitive state to understand what you read and answer questions

Exclusion Criteria:

1. Being currently receiving treatment for known psychological disorders such as depression and anxiety.
2. Having another chronic disease that may cause psychological distress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older, diagnosed with rheumatoid arthritis.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Distress | 10 months
  Presence of distress related with rheumatoid arthritis will be evaluated by Rheumatoid Arthritis Distress Scale.

SECONDARY OUTCOMES:
Disease activity | 10 months
  Disease activity will be evaluated by DAS 28 score.
Functional status | 10 months
  Functional status of patients will be evaluated by HAQ.

CONTACTS AND LOCATIONS:
Overall Officials: Altınay Göksel Karatepe, MD, Principal Investigator — Professor doctor
Locations (1):
- University of Health Sciences Turkey, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matcham F, Rayner L, Steer S, Hotopf M. The prevalence of depression in rheumatoid arthritis: a systematic review and meta-analysis. Rheumatology (Oxford). 2013 Dec;52(12):2136-48. doi: 10.1093/rheumatology/ket169. Epub 2013 Sep 3. PMID 24003249
- [Background] Book K, Marten-Mittag B, Henrich G, Dinkel A, Scheddel P, Sehlen S, Haimerl W, Schulte T, Britzelmeir I, Herschbach P. Distress screening in oncology-evaluation of the Questionnaire on Distress in Cancer Patients-short form (QSC-R10) in a German sample. Psychooncology. 2011 Mar;20(3):287-93. doi: 10.1002/pon.1821. PMID 20669340
- [Background] Woodward S, Dibley L, Coombes S, Bellamy A, Clark C, Czuber-Dochan W, Everelm L, Kutner S, Sturt J, Norton C. Identifying disease-specific distress in patients with inflammatory bowel disease. Br J Nurs. 2016 Jun 23;25(12):649-60. doi: 10.12968/bjon.2016.25.12.649. PMID 27345064
- [Background] Silke L, Kirresh O, Sturt J, Lempp H. Development of the Rheumatoid Arthritis Distress Scale (RADS): a new tool to identify disease-specific distress in patients with Rheumatoid Arthritis. BMC Rheumatol. 2021 Nov 16;5(1):51. doi: 10.1186/s41927-021-00220-4. PMID 34782021